CLINICAL TRIAL: NCT04973345
Title: A Prospective, Blinded, Cross-Over Trial of the Exposure-Response Relationship of Terbutaline Sulfate in Adults With Asthma
Brief Title: Terbutaline Sulfate in Adults With Asthma
Acronym: TBS02
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The TBS02 study was paused indefinitely. No subjects were enrolled or treated, and the study may resume if circumstances change.
Sponsor: Kanecia Obie Zimmerman (Other)
Collaborators: Duke Health (Other); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Kanecia Obie Zimmerman, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00113848; Pro00107910 (Other: Duke site protocol number)
Record Dates: First submitted 2021-07-14; First posted 2021-07-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Terbutaline

STUDY DESIGN:
Intervention Model Description: A Prospective, Blinded, Cross-over Trial of the Exposure-Response Relationship of Terbutaline Sulfate in Adults with Asthma (TBS02)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Terbutaline Arm A (Experimental): • Arm A: (n=6) IV bolus (0.25 mg) over 5 minutes SQ administration (0.25 mg) Participants in Part 1 Arms A and B (n=12) will be randomized to one of two treatment arms.No masking will be applied for Part 1 or for the SQ dosing in Part 2. All IV treatments in Part 2 will be masked, with exception to the unmasked study pharmacist, refer to the MOP for details.
  Interventions: Drug: Terbutaline
- Terbutaline Arm B (Experimental): • Arm B: (n=6) SQ administration (0.25 mg) IV bolus (0.25 mg) over 5 minutes Participants in Part 1 Arms A and B (n=12) will be randomized to one of two treatment arms.No masking will be applied for Part 1 or for the SQ dosing in Part 2. All IV treatments in Part 2 will be masked, with exception to the unmasked study pharmacist, refer to the MOP for details.
  Interventions: Drug: Terbutaline
- Terbutaline Arm C (Experimental): • Arm C: (n=6) SQ (0.25 mg) IV low dose over 5 minutes IV medium dose over 5 minutes IV high dose over 5 minutes Participants in Part 2 (n=18) will be randomized to one of three treatment arms. To maintain masking the first treatment will be 0.25 mg of study drug SQ, followed by one of three IV dose regimes (low, medium, high) below, which are estimated to be 0.1 mg, 0.5 mg, 1.0 mg, but may be adjusted based on the interim analysis completed in Part 1. No masking will be applied for Part 1 or for the SQ dosing in Part 2. All IV treatments in Part 2 will be masked, with exception to the unmasked study pharmacist, refer to the MOP for details.
  Interventions: Drug: Terbutaline
- Terbutaline Arm D (Experimental): • Arm D: (n=6)SQ (0.25 mg) IV medium dose over 5 minutes IV high dose over 5 minutes IV low dose over 5 minutes Participants in Part 2 (n=18) will be randomized to one of three treatment arms. To maintain masking the first treatment will be 0.25 mg of study drug SQ, followed by one of three IV dose regimes (low, medium, high) below, which are estimated to be 0.1 mg, 0.5 mg, 1.0 mg, but may be adjusted based on the interim analysis completed in Part 1. No masking will be applied for Part 1 or for the SQ dosing in Part 2. All IV treatments in Part 2 will be masked, with exception to the unmasked study pharmacist, refer to the MOP for details.
  Interventions: Drug: Terbutaline
- Terbutaline Arm E (Experimental): • Arm E: (n=6) SQ (0.25 mg) IV high dose over 5 minutes IV low dose over 5 minutes IV medium dose over 5 minutes Participants in Part 2 (n=18) will be randomized to one of three treatment arms. To maintain masking the first treatment will be 0.25 mg of study drug SQ, followed by one of three IV dose regimes (low, medium, high) below, which are estimated to be 0.1 mg, 0.5 mg, 1.0 mg, but may be adjusted based on the interim analysis completed in Part 1. No masking will be applied for Part 1 or for the SQ dosing in Part 2. All IV treatments in Part 2 will be masked, with exception to the unmasked study pharmacist, refer to the MOP for details.
  Interventions: Drug: Terbutaline

INTERVENTIONS:
Drug: Terbutaline — management of asthma symptoms

SUMMARY:
The overall aim in Part 1 is to compare the pharmacokinetic (PK)/pharmacodynamics (PD) relationship in intravenous (IV) versus subcutaneous (SQ) terbutaline sulfate to identify the optimal IV dosing range for use in Part 2.

The overall aim in Part 2 is to evaluate the optimal IV dosing of terbutaline sulfate based on PD response and safety data.

DETAILED DESCRIPTION:
Primary Objectives:

1. Describe differences in the PK profiles of terbutaline sulfate administered via the SQ route versus the IV route.
2. Estimate a target plasma concentration and IV dose which achieves maximum FEV1 improvement from baseline and FEV1 AUC.

Secondary Objective: Describe all adverse events (AEs) in participants receiving terbutaline sulfate.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided informed consent
2. History of physician-diagnosed asthma
3. Age ≥18 to <60 at time of consent
4. Past (within 12 months of consent) or current (at screening visit)evidence of airway reactivity, defined as:

   * Documentation of ≥10% FEV1 improvement following bronchodilator OR
   * Positive methacholine challenge (20% or more FEV1 decrease at ≤ 16 mg/mL)
5. Willing and able to undergo study procedures and attend required study visits.
6. Adequate venous access for blood draws and drug administration, as determined by study investigator, or designee
7. Weight ≥ 40kg
8. FEV1 ≥ 60% predicted on day of terbutaline sulfate dosing
9. Systolic blood pressure (BP) ≤ 150 millimeters of Mercury (mmHg) and diastolic BP ≤ 90 mmHg measured after 10 to 15 minutes of rest
10. Heart rate > 45 and < 110 beats per minute (bpm) measured after 10 to 15 minutes of rest
11. Female participants of child-bearing potential: negative pregnancy test (urine hCG) and agreement to use effective contraception (complete abstinence from vaginal intercourse, combination barrier and spermicide, partner vasectomy, bilateral tubal ligation, intrauterine device (IUD), progestin implants, or hormonal) during study participation

Exclusion Criteria:

1. Self-reported pregnancy or lactating or breastfeeding
2. Previous enrollment in the current study (any part)
3. Any chronic respiratory condition besides asthma (including, but not limited to Chronic Obstructive Pulmonary Disease (COPD), emphysema, or interstitial lung disease) that in the opinion of the Principal Investigator (PI) or clinical site investigator, would make the participant unsuitable for the study
4. Body Mass Index (BMI) > 35 kg/m2 (class II or III obesity)
5. Moderate to severe renal impairment, defined as estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2
6. Self-reported combustible cigarette smoking of more than 1 pack per day.
7. Greater than 20 pack-year smoking history
8. Any history of cardiac disease (e.g. coronary insufficiency, cardiac arrhythmias), non-skin cancer, hyperthyroidism, diabetes mellitus type 1, uncontrolled diabetes mellitus type II (HbA1C>7.5 documented within past 12 months of screening) uncontrolled epilepsy (2 or more seizures within the past 12 months and not taking anti-seizure medication)
9. History of ocular, brain, abdominal or thoracic surgery in the 12 months prior to screening
10. Known hypersensitivity to terbutaline sulfate or albuterol
11. Use of any medications from the following classes within 28 days prior to Visit 1: monoamine oxidase inhibitors, tricyclic antidepressants, beta blockers, non-potassium-sparing antihypertensive diuretics, or systemic corticosteroids
12. Self-reported respiratory tract infection in the 14 days prior to Visit 1
13. Any current chronic condition or past history of disease that, in the opinion of the PI would make the participant unsuitable for the study
14. Baseline prolongation of QTc (QTc ≥ 460 ms by Fridericia's formula)
15. Participation in another research study that includes use of any investigational drug treatment within the 30 days prior to Visit 1, or planned participation during the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PK: Maximum concentration (CMAX) | 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, and next calendar day after dose
  Describe differences in the PK profiles of terbutaline sulfate administered via the SQ route versus the IV route.
PK: Time to Research Maximum Concentration (Tmax) | 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours after dose
  Describe differences in the PK profiles of terbutaline sulfate administered via the SQ route versus the IV route.
PK: Clearance (Cl) | 5 mins, 15 mins, 30 mins, 45 mins, 1 hr, 2 hrs, 3 hrs, 4 hrs, 6 hrs, after dose
  Describe differences in the PK profiles of terbutaline sulfate administered via the SQ route
PK: Volume of Distribution (Vd) | 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours after dose
  Describe differences in the PK profiles of terbutaline sulfate administered via the SQ route
PK: Half Life (t1/2) | 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours after dose
  Describe differences in the PK profiles of terbutaline sulfate administered via the SQ route
Concentration Achieving Maximum FEV1 Improvement (CeMax) | 0-6 hours
  Estimate a target plasma concentration and IV dose which achieves maximum FEV1 improvement from baseline and FEV1 AUC 0 to 6 hours.
Area Under the Concentration Time Curve (AUC) | 5 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, and next calendar day after dose
  Describe differences in the PK profiles of terbutaline sulfate administered via the SQ route versus the IV route.
Forced Expiratory Volume in 1 second (FEV1) | 0-6 hours
  Estimate a target plasma concentration and IV dose which achieves maximum FEV1 improvement from baseline and FEV1 AUC 0 to 6 hours.

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | From baseline through the end of study (Part I up to 60 days, Part II up to 180 days)
  Adverse events (AEs) in participants receiving terbutaline sulfate.
Number of Serious Adverse Events (SAEs) | From baseline through the end of study (Part I up to 60 days, Part II up to 180 days)
  Serious Adverse Events (SAEs) in participants receiving terbutaline sulfate.
Number of Suspected Unexpected Serious Adverse Reactions (SUSARs) | From baseline through the end of study (Part I up to 60 days, Part II up to 180 days)
  Suspected Unexpected Serious Adverse Reactions (SUSARs) in participants receiving terbutaline sulfate.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lang, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - University of Colorado, Aurora, Colorado
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT04973345/ICF_000.pdf